CLINICAL TRIAL: NCT05858580
Title: Pilot Study of a Home-based Program to Promote Healthy Diet and Activity in Rural-dwelling Children
Brief Title: The Bennett Kids PowerUP Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00100266; 40010049 (Other: American Diabetes Association)
Record Dates: First submitted 2023-03-16; First posted 2023-05-15 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Childhood; Type2diabetes
Keywords: Rural Population; Child Health; Physical Activity; Healthy Diet; Veggie Meter; Family-based Approach
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 in blocks of 6 to the intervention or control groups with the Randomization Module of the Research Data Capture (REDCap).
Who Masked: Outcomes Assessor
Masking Description: Data collectors will be blinded to the participant's assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention participants will receive approximately 25 hours of programming (over a 6-month period) related to the promotion of physical activity and healthy diet through:
  1. 16 self-contained, parent-guided activity kits,
  2. 9 one-on-one health coach/support sessions in-person or virtual by a trained health coach,
  3. unlimited access to a resource toolbox.
  Interventions: Behavioral: Bennett Kids PowerUP Project
- Control Group (No Intervention): Control group programming consists of:
  1. 6 parent-guided activity kits focused on STEM activities,
  2. 6 monthly check-in calls to support retention.
  The investigators will use Home Science Lab STEM kits designed for English- and Spanish-speaking children aged 6-11 years. The STEM kits do not include any physical health content. Kits will be mailed monthly to the participants' home. To maximize retention in the control group, staff will contact participants each month to confirm the kit was received, encourage completion of the kits, ask about their experience, and answer questions.

INTERVENTIONS:
Behavioral: Bennett Kids PowerUP Project — Information targeting dietary and activity behaviors while also identifying and addressing barriers to permanent lifestyle change. The foundation of the curriculum is the Diabetes Prevention Program Lifestyle Balance and its subsequent adaptations for non-Native adult, Native adult, and Native child populations.
  Arms: Intervention Group

SUMMARY:
The study proposes a randomized pilot and feasibility study of a lifestyle modification program to promote healthy diet and activity in rural-dwelling children to reduce Type 2 Diabetes risks.

Intervention participants will receive 6 months of programming to include:

* 16 activity packs;
* 9 health coach sessions;
* unlimited access to a resource toolbox.

Control participants will receive 6 activity packs promoting science, technology, engineering, and math (STEM) learning and 6 check-in calls to support retention.

DETAILED DESCRIPTION:
The rising prevalence of obesity and type 2 diabetes (T2D) at increasingly younger ages compels development of new strategies to combat these preventable conditions. Healthy diet and activity are critical to reducing risk, yet these behaviors decline starting in childhood. These trends are most troubling in rural areas, where youth consume more calories and sugar-sweetened beverages but less fruit and whole grains; engage in less physical activity; and are more likely to have overweight or obesity than urban peers. Given unhealthy behaviors are set by adolescence, promoting healthy diet and activity in rural children is crucial to reducing rural-urban disparities in obesity and T2D across the lifecourse.

The investigators have developed a multi-component, family-based intervention to improve diet and activity in children at risk of youth-onset obesity and T2D. The pilot study will gather necessary and sufficient data on feasibility, acceptability, and effect size to finalize the design of a clinical trial.

The investigators will recruit 60 English- or Spanish-speaking children in 2nd to 5th grades from rural communities in Colorado or North Carolina. Participants will be randomized to 6 months of intervention or control programming. Intervention participants will receive approximately 25 hours of programming over 6 months through a) 16 self-contained, parent-guided activity kits, b) 9 one-on-one health coach/support sessions in-person or virtual by a trained health coach, and c) unlimited access to a resource toolbox. Control participants will receive 6 activity kits promoting science, technology, engineering, and math (STEM) learning and will receive 6 check-in calls to support retention.

Standardized measures will be collected at 0 and 7 months. Qualitative interviews will also be conducted at 7 months. Process measures will be tracked by staff throughout the study. With positive results, this innovative pilot study will form the foundation of a clinical trial to evaluate the sustained impact of an at-home, family-based intervention to promote diet and activity in rural children, which can subsequently be disseminated and implemented among the 13 million children living in rural US settings and reduce T2D risks.

ELIGIBILITY:
Inclusion Criteria:

* 7-to-10-years-old
* Living in rural Colorado or rural North Carolina
* English- or Spanish-speaking
* Has 1 parent or primary caregiver willing to actively participate

Exclusion Criteria:

* Medical diagnosis of diabetes
* Serious child or parent health concerns that would interfere with participation
* Plans to move out of the area during the study period
* Lives with another child who previously participated in the study

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Dietary Intake (MyPyramid Equivalents) at 7 months | Month 7
  Diet will be assessed with 24-hour dietary recalls using the Automated Self Administered system (ASA24). This system uses the USDA multiple-pass method to query all foods and supplements consumed in the prior 24 hours and produces daily and individual food estimates for macronutrients, micronutrients, and MyPyramid Equivalents (such as servings of vegetables, fruits, whole grains, solid fats, and added sugars).
Change in Fruit and Vegetable Intake (carotenoid concentration) at 7 months | Month 7
  Use the Veggie Meter (Longevity Link, Salt Lake City, UT) to assess carotenoids, a biomarker of fruit and vegetable intake. The device estimates total dermal carotenoid concentration by illuminating the fingertip with a blue wavelength laser light and detecting vibrational/rotational energy levels of molecules, correcting for hemoglobin and melanin levels.
Change in Sugar-Sweetened Beverage Intake (carbon isotope ratio) at 7 months | Month 7
  Collect red blood cells to measure the carbon isotope ratio, a biomarker of sugar-sweetened beverage intake. Samples will be analyzed via continuous-flow isotope ratio mass spectrometry at the University of Alaska Stable Isotope Facility.

SECONDARY OUTCOMES:
Change in Physical Activity at 7 months | Month 7
  7-day accelerometry using the wGT3X-BT water resistant tri-axial accelerometer (Actigraph LLC, Pensacola, FL). Monitors are worn on an elastic band on the waist for 7 days. Recordings with greater than or equal to 10 hours of data on 4 or more days will be coded using established youth cut-points to determine the daily minutes of moderate-vigorous activity and sedentary time.
Change in Screen Time at 7 months | Month 7
  CommonSense Media Use Survey to estimate minutes/day across relevant categories (e.g. recreational use vs communication vs educational). Our screen time analyses will focus on recreational screen time but also report on the other types.

OTHER OUTCOMES:
Change in Glucose levels at 7 months | Month 7
  Fasting serum samples analysis (Hexokinase, UV)
Change in Insulin values at 7 months | Month 7
  Fasting serum samples analysis (chemiluminescence immunoassay)
Change in Body Mass Index (BMI) values at 7 months | Month 7
  Measured height, weight - Under 18.5 - you are very underweight and possibly malnourished. 18.5 to 24.9 - you have a healthy weight range for young and middle-aged adults. 25.0 to 29.9 - you are overweight. Over 30 - you are obese.
Program Engagement | Month 7
  Number of activity kits completed
Completion of coaching sessions | Month 7
  Number of health coach sessions completed
Use of toolbox number | Month 7
  Report on frequency of use of the resource toolbox
Process Measures | Month 7
  Staff records of the actual schedule (order and timing) of mailed activity kits and health coach sessions
Acceptability and Engagement Barriers | Month 7
  Semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Sauder, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No